CLINICAL TRIAL: NCT07182188
Title: Post-Market Application Study and Efficacy/Safety Evaluation of a Vascular Interventional Robotic System for Cerebral Angiography: A Multicenter Randomized Controlled Trial
Brief Title: A Clinical Trial of Vascular Interventional Robotic System for Cerebral Angiography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuanli Zhao, Director of the Department of Neurosurgery, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MR-11-24-024538
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Crerbral Angiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Manual Endovascular Angiography (No Intervention)
- Vascular Interventional Robotic System Assisted Angiography (Experimental)
  Interventions: Device: Vascular Interventional Robotic System

INTERVENTIONS:
Device: Vascular Interventional Robotic System — The cerebral angiography will be performed by using the vascular interventional robotic system
  Arms: Vascular Interventional Robotic System Assisted Angiography

SUMMARY:
This study aims to conduct a post-market, multicenter clinical trial utilizing an interventional robotic system for cerebral angiography. By comparing it with traditional angiography procedures, the study will systematically evaluate the efficacy and safety of robot-assisted angiography in real clinical settings. Researchers will compare the ordinary angiography to assess the clinical success rate, operation time, radiation absorption, complication rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years;
2. Suspected vascular lesions in the head and neck, or other conditions involving head and neck vessels requiring whole-brain angiography for definitive diagnosis or to aid treatment decisions. Including but not limited to: intracranial aneurysms, arteriovenous malformations, cavernous malformations, arteriovenous fistulas, Moyamoya disease, Moyamoya syndrome, subarachnoid hemorrhage, symptomatic intracranial artery stenosis/occlusion, stenosis/occlusion of the carotid/subclavian/vertebral arteries, acute/ chronic subdural hematoma, etc;
3. American Society of Anesthesiologists (ASA) physical status classification I-III (no severe cardiopulmonary dysfunction);
4. Patients who voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients who are to undergo surgery at the same time as cerebral angiography;
2. Renal dysfunction (serum creatinine > 133 μmol/L or estimated glomerular filtration rate < 60 mL/min/1.73 m²);
3. Patients with known allergy to iodinated contrast media;
4. Coagulation disorders (prothrombin time >16s, activated partial thromboplastin time >45s, or platelet count <100×10⁹/L);
5. Severe infection, skin ulceration, or vascular anatomical abnormalities at the puncture site (e.g., bilateral femoral artery occlusion);
6. Pregnant or lactating women;
7. Patients with severe cognitive impairment;
8. Patients with psychiatric disorders;
9. Patients unable to undergo head magnetic resonance imaging (MRI), e.g., those with metallic implants, claustrophobia, or other contraindications;
10. Patients with other severe advanced or terminal illnesses;
11. Patients currently participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Angiography Success Rate | At the end of surgery
  Assessment of the success rate of the surgeon in completing cerebral angiography examination through the operation of vascular interventional robotic system or manual way.
Complication Rate | At the day after surgery
  Potential complications include: ① Directly related to the interventional procedure: Vascular injury (vessel rupture, perforation, spasm, gas embolism, and thrombosis); ② Neurological complications: New-onset neurological deficits (transient/permanent), new-onset cerebral ischemia, or new-onset intracerebral hemorrhage, confirmed by postoperative imaging; ③ Systemic complications: Cardiac events, gastrointestinal bleeding, renal dysfunction, etc.

SECONDARY OUTCOMES:
Operation Time | At the end of surgery
  Record and compare the duration of each surgical procedure.
Super-selective Success Rate | At the end of surgery
  Assessing the success rate of the surgeon in performing super-selective catheterization of each cerebral vessels through the operation of vascular interventional robotic system or manual way.
Super-selective Catheterization Time for Vessels | At the end of surgery
  Calculate and compare the average time taken for surgeon to perform super-selective catheterization for each target vessel during each surgical procedure.
Digital Subtraction Angiography (DSA) Fluoroscopy Time | At the end of surgery
  Calculate and compare the average time of fluoroscopy during cerebral angiography for each surgical procedure.
Primary Operator Radiation Absorbed Dose | At the end of surgery
  Record and compare the absorbed dose of radiation received by the primary operator during each surgical procedure.
Participant Radiation Absorbed Dose | At the end of surgery
  Record and compare the absorbed dose of radiation received by the participant during each surgical procedure.
Vascular Interventional Robotic System Performance Evaluation | At the end of surgery
  The surgical physician rate a score (0-10) after the surgery to subjectively evaluate the performance of the vascular interventional robotic system during the angiographic examination procedure.
Frequence of robotic operations transition to manual operations | At the end of surgery
  Document the frequence where robotic operations transition to manual operations due to certain force majeure events.
Operation Preparation Time | At the end of Surgery
  Calculate and compare the time from when participants enter the operating room until the primary operator formal start the surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No
The vascular interventional robotic system includes proprietary technical features that are integral to the IPD. Publicly sharing IPD would inadvertently disclose proprietary information, which could compromise the manufacturer's intellectual property rights and hinder future development of the technology for broader clinical use.

REFERENCES:
- [Background] Liu H, Li C, Ren S, Li T, Zhong H, Jia J, Yang H, Qi Y, Feng J, Li Y, Wang Y. Efficacy and safety of a neurointerventional operation robotic assistance system in cerebral angiography. Stroke Vasc Neurol. 2024 Jun 21;9(3):243-251. doi: 10.1136/svn-2022-002260. PMID 37612055
- [Background] Zhang Y, Xu H, Sun J, Chen WH, Zhang Y, Chen M, Yi T, Wu YM, Cheng G, Guo J, Yang P, Guo S, Liu J. Safety and efficacy of cerebral robot assisted angiography: randomized comparison of robotic versus manual procedures. J Neurointerv Surg. 2025 Jul 9:jnis-2025-023412. doi: 10.1136/jnis-2025-023412. Online ahead of print. PMID 40633938
- [Background] Beaman C, Gautam A, Peterson C, Kaneko N, Ponce L, Saber H, Khatibi K, Morales J, Kimball D, Lipovac JR, Narsinh KH, Baker A, Caton MT, Smith ER, Nour M, Szeder V, Jahan R, Colby GP, Cord BJ, Cooke DL, Tateshima S, Duckwiler G, Waldau B; Robotics Working Group; Robotic Working Group. Robotic Diagnostic Cerebral Angiography: A Multicenter Experience of 113 Patients. J Neurointerv Surg. 2024 Jun 17;16(7):726-730. doi: 10.1136/jnis-2023-020448. PMID 37468266